CLINICAL TRIAL: NCT01461538
Title: A Phase 2, Open-label Study of Brentuximab Vedotin in Patients With CD30-positive Nonlymphomatous Malignancies
Brief Title: Brentuximab Vedotin in Patients With CD30-positive Nonlymphomatous Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGN35-013
Record Dates: First submitted 2011-10-24; First posted 2011-10-28 (Estimated); Results first posted 2016-03-04 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-02

CONDITIONS: Acute Lymphoid Leukemia; Acute Myeloid Leukemia; Anemia, Refractory, With Excess of Blasts; Solid Tumors
Keywords: Acute Lymphoid Leukemia; Myelodysplastic Syndrome; Acute Myeloid Leukemia; Solid Tumors; Anemia, Refractory, with Excess of Blasts; Antibodies, Monoclonal; Antibody-Drug Conjugate; Antigens, CD30; Drug Therapy; Hematologic Diseases; Immunotherapy; Monomethyl Auristatin E
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts; Myelodysplastic Syndromes; Hematologic Diseases | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Brentuximab vedotin 1.8 mg/kg (Experimental): Brentuximab vedotin 1.8 mg/kg every 3 weeks by IV infusion
  Interventions: Drug: brentuximab vedotin
- Brentuximab vedotin 2.4 mg/kg (Experimental): Brentuximab vedotin 2.4 mg/kg every 3 weeks by IV infusion
  Interventions: Drug: brentuximab vedotin
- Brentuximab vedotin 1.2 mg/kg (Experimental): Brentuximab vedotin 1.2 mg/kg weekly, 3 out of 4 weeks, by IV infusion
  Interventions: Drug: brentuximab vedotin

INTERVENTIONS:
Drug: brentuximab vedotin — 1.8 mg/kg every 3 weeks by intravenous (IV) infusion
  Other Names: Adcetris; SGN-35
  Arms: Brentuximab vedotin 1.8 mg/kg
Drug: brentuximab vedotin — 2.4 mg/kg every 3 weeks by intravenous (IV) infusion
  Other Names: Adcetris; SGN-35
  Arms: Brentuximab vedotin 2.4 mg/kg
Drug: brentuximab vedotin — 1.2 mg/kg weekly, 3 out of 4 weeks, by intravenous (IV) infusion
  Other Names: Adcetris; SGN-35
  Arms: Brentuximab vedotin 1.2 mg/kg

SUMMARY:
This is an open-label, multicenter, phase 2 clinical trial to evaluate the antitumor activity of brentuximab vedotin as a single agent in patients with CD30-positive nonlymphomatous malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed by central review CD30-positive nonlymphomatous malignancy
* Have failed, refused, or have been deemed ineligible for standard therapy
* Measurable disease
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1 or a Karnofsky or Lansky Performance Status score greater than or equal to 70

Exclusion Criteria:

* Primary diagnosis of lymphoma or central nervous system (CNS) malignancy
* History of another primary invasive malignancy that has not been definitively treated or in remission for at least 3 years
* Evidence of active cerebral/meningeal disease

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2011-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Josephson, MD, Study Director — Seagen Inc.
Locations (29):
- United States (29):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope, Duarte, California
  - PMK Medical Group Inc., DBA Ventura County Hematology Oncology Specialists, Oxnard, California
  - Rocky Mountain Cancer Centers - Aurora, Aurora, Colorado
  - Mayo Clinic Cancer Center, Jacksonville, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Minnesota Oncology Hematology P.A., Minneapolis, Minnesota
  - New York Oncology Hematology, P.C., Albany, New York
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Willamette Valley Cancer and Research / USOR, Eugene, Oregon
  - Northwest Cancer Specialists, P.C., Tulatin, Oregon
  - St. Francis Hospital, Greenville, South Carolina
  - Texas Oncology - Bedford, Bedford, Texas
  - Texas Oncology - Medical City Dallas, Dallas, Texas
  - Texas Oncology - Dallas Presbyterian, Dallas, Texas
  - Texas Oncology Denton South, Denton, Texas
  - Texas Oncology - Fort Worth 12th Avenue, Fort Worth, Texas
  - MD Anderson Cancer Center / University of Texas, Houston, Texas
  - MD Anderson Cancer Center Leukemia Group, Houston, Texas
  - Texas Oncology - Central Austin Cancer Center, Round Rock, Texas
  - Cancer Centers of South Texas - HOAST, San Antonio, Texas
  - Texas Oncology - Waco, Waco, Texas
  - Oncology and Hematology Assoc of SW VA DBA Blue Ridge Cancer Care, Blacksburg, Virginia
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Puget Sound Cancer Centers, Edmonds, Washington
  - Cancer Care Northwest, Spokane Valley, Washington
  - Yakima Valley Memorial Hospital / North Star Lodge, Yakima, Washington

REFERENCES:
- [Derived] Albany C, Einhorn L, Garbo L, Boyd T, Josephson N, Feldman DR. Treatment of CD30-Expressing Germ Cell Tumors and Sex Cord Stromal Tumors with Brentuximab Vedotin: Identification and Report of Seven Cases. Oncologist. 2018 Mar;23(3):316-323. doi: 10.1634/theoncologist.2017-0544. Epub 2017 Dec 8. PMID 29222199
- [Derived] Borate U, Mehta A, Reddy V, Tsai M, Josephson N, Schnadig I. Treatment of CD30-positive systemic mastocytosis with brentuximab vedotin. Leuk Res. 2016 May;44:25-31. doi: 10.1016/j.leukres.2016.02.010. Epub 2016 Feb 27. PMID 26994848
- [Derived] Giannatempo P, Paolini B, Miceli R, Raggi D, Nicolai N, Fare E, Catanzaro M, Biasoni D, Torelli T, Stagni S, Piva L, Mariani L, Salvioni R, Colecchia M, Gianni AM, Necchi A. Persistent CD30 expression by embryonal carcinoma in the treatment time course: prognostic significance of a worthwhile target for personalized treatment. J Urol. 2013 Nov;190(5):1919-24. doi: 10.1016/j.juro.2013.04.057. Epub 2013 Apr 25. PMID 23624209

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Oct 2011 - Dec 2014
Pre-assignment Details: One additional patient enrolled, but withdrew prior to treatment group assignment.
Groups:
- BV 1.8 mg/kg Q3Week: Brentuximab vedotin 1.8 mg/kg every 3 weeks by intravenous (IV) infusion in patients with CD30-positive solid tumors or leukemia
- BV 2.4 mg/kg Q3Week: Brentuximab vedotin 2.4 mg/kg every 3 weeks by intravenous (IV) infusion in patients with CD30-positive solid tumors or leukemia
- BV 1.2 mg/kg Q1Week: Brentuximab vedotin 1.2 mg/kg weekly, 3 out of 4 weeks, by intravenous (IV) infusion in patients with acute leukemia or myelodysplastic syndrome (MDS)
Period: Overall Study
Arm/Group | BV 1.8 mg/kg Q3Week | BV 2.4 mg/kg Q3Week | BV 1.2 mg/kg Q1Week
Started | 46 | 28 | 9
Completed | 28 | 20 | 7
Not Completed | 18 | 8 | 2
Not completed — Death | 15 | 6 | 2
Not completed — Study Stopped by Sponsor | 2 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received treatment. One additional patient enrolled, but withdrew prior to treatment group assignment.
Groups:
- Total: Total of all reporting groups
Arm/Group | BV 1.8 mg/kg Q3Week | BV 2.4 mg/kg Q3Week | BV 1.2 mg/kg Q1Week | Total
Number analyzed (Participants) | 46 | 28 | 9 | 83
Age, Continuous [Median (Full Range); unit: years] | 64 [24 to 85] | 64 [18 to 85] | 76 [33 to 87] | 65 [18 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 12 | 4 | 37
  Male | 25 | 16 | 5 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 0 | 4
  Not Hispanic or Latino | 44 | 26 | 9 | 79
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 2
  White | 42 | 25 | 9 | 76
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 46 | 28 | 9 | 83
Eastern Cooperative Oncology Group Performance Status [Number; unit: participants] — 0 = Normal activity; 1 = Symptoms but ambulatory; 2 = In bed <50% of the time; 3 = In bed >50% of the time; 4 = 100% bedridden; 5 = Dead
  participants
    0 | 13 | 5 | 1 | 19
    1 | 20 | 15 | 5 | 40
    2 | 0 | 0 | 1 | 1
    3-5 | 0 | 0 | 0 | 0
    Missing | 13 | 8 | 2 | 23
Height [Median (Full Range); unit: centimeters (cm)] | 170.2 [142 to 188] | 171.9 [150 to 186] | 167.6 [144 to 180] | 170.2 [142 to 188]
Weight [Median (Full Range); unit: kilograms (kg)] | 74.8 [46 to 109] | 75.1 [49 to 104] | 73.4 [45 to 137] | 74.8 [45 to 137]
Body Mass Index [Median (Full Range); unit: kg per meter squared (kg/m^2)] | 25.3 [19 to 40] | 27.4 [18 to 36] | 26.3 [20 to 47] | 26.0 [18 to 47]

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) by Investigator
Description: Percentage of participants who achieved a best response of complete response/remission (CR), CR without hematologic recovery (CRi; leukemia only), or partial remission (PR) per the applicable response criteria. Response criteria for solid tumors (by radiographic tumor imaging) per Response Evaluation Criteria for Solid Tumors (RECIST) 1.1 (Eisenhauer 2009); response criteria for leukemia (by peripheral blood and bone marrow aspirate or biopsy) per International Working Group (Cheson 2003).
Time Frame: Up to approximately 3 years
Population: Efficacy-evaluable population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Solid Tumors: Participants with solid tumors
- Leukemia: Participants with acute leukemia or high grade MDS (refractory anemia with excess blasts-2)
Arm/Group | Solid Tumors | Leukemia
Number analyzed (Participants) | 59 | 14
percentage of participants | 12 [4.9 to 22.9] | 14 [1.8 to 42.8]

2. Secondary Outcome: Complete Remission (CR) Rate by Investigator
Description: Percentage of participants who achieved a best response of CR per the applicable response criteria. Response criteria for solid tumors (by radiographic tumor imaging) per Response Evaluation Criteria for Solid Tumors (RECIST) 1.1 (Eisenhauer 2009); response criteria for leukemia (by peripheral blood and bone marrow aspirate or biopsy) per International Working Group (Cheson 2003).
Time Frame: Up to approximately 3 years
Population: Efficacy-evaluable population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Solid Tumors | Leukemia
Number analyzed (Participants) | 59 | 14
percentage of participants | 2 [0.0 to 9.1] | 0 [0 to 23.2]

3. Secondary Outcome: Duration of Objective Response by Kaplan-Meier Analysis
Description: Duration of objective response (CR [+CRi; leukemia] + PR), defined as time of initial response until disease progression or death. Response criteria for solid tumors (by radiographic tumor imaging) per Response Evaluation Criteria for Solid Tumors (RECIST) 1.1 (Eisenhauer 2009); response criteria for leukemia (by peripheral blood and bone marrow aspirate or biopsy) per International Working Group (Cheson 2003).
Time Frame: Up to approximately 2 years
Population: Participants with objective response (CR [+CRi; leukemia] + PR)
Measure: Median (Full Range); unit: months
Arm/Group | Solid Tumors | Leukemia
Number analyzed (Participants) | 7 | 2
months | 2.9 [1.5 to 23.5] | 2.1 [1.0 to 3.1]

4. Secondary Outcome: Duration of Complete Response by Kaplan-Meier Analysis
Description: Duration of CR, defined as time of initial response until disease progression or death. Response criteria for solid tumors (by radiographic tumor imaging) per Response Evaluation Criteria for Solid Tumors (RECIST) 1.1 (Eisenhauer 2009); response criteria for leukemia (by peripheral blood and bone marrow aspirate or biopsy) per International Working Group (Cheson 2003).
Time Frame: Up to approximately 2 years
Population: Participants with CR
Measure: Median (Full Range); unit: months
Arm/Group | Solid Tumors | Leukemia
Number analyzed (Participants) | 1 | 0
months | 22.3 [22.3 to 22.3] |

5. Secondary Outcome: Progression-Free Survival by Kaplan-Meier Analysis
Description: Progression-free survival, defined as time from start of study treatment to disease progression per investigator or death due to any cause
Time Frame: Up to approximately 2 years
Population: All treated patients, excluding 3 patients without available response results
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Solid Tumors | Leukemia
Number analyzed (Participants) | 63 | 17
months | 2.1 [1.3 to 2.8] | 0.7 [0.7 to 1.3]

6. Secondary Outcome: Adverse Events by Severity, Seriousness, and Relationship to Treatment
Description: Counts of participants who had treatment-emergent adverse events (TEAE, defined as newly occurring or worsening after first dose on Study SGN35-013). Serious adverse events are reported from the time of informed consent. National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE version 4.03) were used to assess severity (1=mild, 2=moderate, 3=severe, 4=life-threatening/disabling, 5=fatal). Relatedness to study drug was assessed by the investigator (Yes/No). Participants with multiple occurrences of an adverse event within a category are counted once within the category.
Time Frame: Up to approximately 3 years
Population: All treated patients
Measure: Number; unit: participants
Arm/Group | BV 1.8 mg/kg Q3Week | BV 2.4 mg/kg Q3Week | BV 1.2 mg/kg Q1Week
Number analyzed (Participants) | 46 | 28 | 9
participants
  Any TEAE | 45 | 28 | 9
  TEAE related to study drug | 31 | 24 | 5
  TEAE with severity grade >/=3 | 31 | 18 | 7
  Discontinued treatment due to adverse event | 5 | 2 | 2
  Serious adverse event | 24 | 13 | 5
  Serious adverse event related to study drug | 5 | 6 | 2
  Deaths (within 30 days of last dose) | 10 | 6 | 2

7. Secondary Outcome: Laboratory Abnormalities >/= Grade 3
Description: Counts of study participants with post-baseline laboratory abnormalities of Grade 3 or greater per NCI CTCAE version 4.03. Participants with multiple occurrences of a laboratory abnormality within a category are counted once in that category
Time Frame: Up to approximately 3 years
Population: All treated patients
Measure: Number; unit: participants
Arm/Group | BV 1.8 mg/kg Q3Week | BV 2.4 mg/kg Q3Week | BV 1.2 mg/kg Q1Week
Number analyzed (Participants) | 46 | 28 | 9
participants
  Any >/= Grade 3 laboratory abnormality | 24 | 12 | 9
  Alanine aminotransferase high | 0 | 1 | 1
  Albumin low | 2 | 3 | 0
  Alkaline phosphatase high | 0 | 1 | 0
  Aspartate aminotransferase high | 0 | 1 | 0
  Bilirubin high | 0 | 1 | 0
  Calcium low | 1 | 1 | 0
  Glucose high | 2 | 1 | 0
  Glucose low | 1 | 0 | 0
  Sodium low | 4 | 2 | 0
  Urate high | 2 | 0 | 0
  Prothrombin INR high | 0 | 0 | 1
  Absolute neutrophil count low | 6 | 2 | 5
  Hemoglobin low | 4 | 0 | 3
  Leukocytes high | 0 | 1 | 1
  Leukocytes low | 4 | 0 | 4
  Lymphocytes high | 1 | 2 | 0
  Lymphocytes low | 9 | 3 | 1
  Neutrophils low | 6 | 3 | 7
  Platelets low | 4 | 4 | 7

8. Secondary Outcome: Brentuximab Vedotin Antibody-Drug Conjugate (ADC) Concentration at End of Infusion (Ceoi)
Time Frame: Up to approximately 3 years
Population: All treated patients with available ADC Ceoi results
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | BV 1.8 mg/kg Q3Week | BV 2.4 mg/kg Q3Week | BV 1.2 mg/kg Q1Week
Number analyzed (Participants) | 42 | 25 | 9
ug/mL | 40 (26) | 54 (28) | 25 (23)

9. Secondary Outcome: Brentuximab Vedotin Antibody-Drug Conjugate (ADC) Trough Concentration (Ctrough)
Time Frame: Up to approximately 3 years
Population: All treated patients with available ADC Ctrough results
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | BV 1.8 mg/kg Q3Week | BV 2.4 mg/kg Q3Week | BV 1.2 mg/kg Q1Week
Number analyzed (Participants) | 34 | 10 | 9
ug/mL | 0.36 (180) | 0.55 (210) | 1.5 (48)

10. Secondary Outcome: Maximum Concentration (Cmax) of Brentuximab Vedotin Monomethyl Auristatin E (MMAE)
Time Frame: Up to approximately 3 years
Population: All treated patients with available Cmax of MMAE results
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | BV 1.8 mg/kg Q3Week | BV 2.4 mg/kg Q3Week | BV 1.2 mg/kg Q1Week
Number analyzed (Participants) | 43 | 25 | 9
ng/mL | 4.0 (78) | 6.2 (71) | 2.6 (83)

11. Secondary Outcome: Brentuximab Vedotin Monomethyl Auristatin E (MMAE) Trough Concentration (Ctrough)
Time Frame: Up to approximately 3 years
Population: All treated patients with available MMAE Ctrough results
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | BV 1.8 mg/kg Q3Week | BV 2.4 mg/kg Q3Week | BV 1.2 mg/kg Q1Week
Number analyzed (Participants) | 34 | 11 | 9
ng/mL | 0.22 (92) | 0.35 (82) | 1.5 (65)

12. Secondary Outcome: Incidence of Anti-therapeutic Antibodies (ATA)
Description: Counts of participants with post-baseline anti-brentuximab vedotin antibodies. Persistently positive is defined as confirmed ATA in more than 2 post-baseline samples and transiently positive is defined as confirmed ATA in 1 or 2 post-baseline samples.
Time Frame: Up to approximately 3 years
Population: Immunogenicity-evaluable set
Measure: Number; unit: participants
Arm/Group | BV 1.8 mg/kg Q3Week | BV 2.4 mg/kg Q3Week | BV 1.2 mg/kg Q1Week
Number analyzed (Participants) | 36 | 23 | 8
participants
  Baseline (BL) negative | 33 | 21 | 8
  BL negative, negative post-BL | 14 | 14 | 8
  BL negative, transiently positive post-BL | 18 | 6 | 0
  BL negative, persistently positive post-BL | 1 | 1 | 0
  BL positive | 3 | 2 | 0
  BL positive, negative post-BL | 1 | 0 | 0
  BL positive, transiently positive post-BL | 2 | 1 | 0
  BL positive, persistently positive post-BL | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 3 years
Description: TEAEs, defined as newly occurring (not present at baseline) or worsening after first dose of brentuximab vedotin
Arm/Group | BV 1.8 mg/kg Q3Week | BV 2.4 mg/kg Q3Week | BV 1.2 mg/kg Q1Week
Serious Adverse Events (participants affected / at risk) | 24/46 | 13/28 | 5/9
Other Adverse Events (participants affected / at risk) | 42/46 | 28/28 | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BV 1.8 mg/kg Q3Week (N=46) | BV 2.4 mg/kg Q3Week (N=28) | BV 1.2 mg/kg Q1Week (N=9)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Systemic mastocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0
Pyrexia (General disorders) | 1 | 1 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1
Hepatosplenomegaly (Hepatobiliary disorders) | 0 | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 1
Sepsis (Infections and infestations) | 3 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 2 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Acute myeloid leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1
Erythroleukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Rhabdomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 0
Azotemia (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BV 1.8 mg/kg Q3Week (N=46) | BV 2.4 mg/kg Q3Week (N=28) | BV 1.2 mg/kg Q1Week (N=9)
Anemia (Blood and lymphatic system disorders) | 6 | 1 | 4
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 3 | 1
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 3
Sinus tachycardia (Cardiac disorders) | 1 | 2 | 1
Tachycardia (Cardiac disorders) | 3 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 3 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 3 | 0
Ascites (Gastrointestinal disorders) | 3 | 2 | 0
Constipation (Gastrointestinal disorders) | 9 | 7 | 1
Diarrhea (Gastrointestinal disorders) | 14 | 5 | 2
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 13 | 11 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 11 | 7 | 0
Asthenia (General disorders) | 4 | 0 | 0
Chest pain (General disorders) | 1 | 2 | 0
Chills (General disorders) | 6 | 2 | 1
Fatigue (General disorders) | 26 | 10 | 3
Malaise (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 2 | 0
Edema peripheral (General disorders) | 4 | 6 | 1
Pain (General disorders) | 2 | 0 | 2
Pyrexia (General disorders) | 6 | 4 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 3 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 1
Weight decreased (Investigations) | 2 | 4 | 0
Decreased appetite (Metabolism and nutrition disorders) | 11 | 9 | 2
Dehydration (Metabolism and nutrition disorders) | 4 | 3 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 3 | 4 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 3 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 5 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 5 | 4 | 0
Headache (Nervous system disorders) | 5 | 3 | 0
Peripheral motor neuropathy (Nervous system disorders) | 5 | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 8 | 7 | 1
Anxiety (Psychiatric disorders) | 4 | 2 | 0
Delirium (Psychiatric disorders) | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 3 | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 6 | 3
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 7 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 7 | 1
Rash (Skin and subcutaneous tissue disorders) | 8 | 4 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 3 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Flushing (Vascular disorders) | 1 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days